CLINICAL TRIAL: NCT05661734
Title: A Phase 3, Single-arm Study Evaluating the Safety and Effectiveness of VX-548 for Acute Pain
Brief Title: A Single-arm Study to Evaluate Safety and Effectiveness of VX-548 for Acute Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX22-548-107
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Suzetrigine (SUZ) (Experimental): Participants received SUZ 100 milligram (mg) as first dose, followed by SUZ 50 mg every 12 hours (q12h) for 14 days or until pain resolves, whichever occurs first.
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: Suzetrigine — Tablets for oral administration.
  Other Names: VX-548; SUZ

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of VX-548 in treating acute pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of greater than or equal to (≥) 18.0 to less than (<) 40.0 kilogram per meter square (kg/m^2)
* Non-surgical participants with pain of new origin (not related to a prior known condition) that is moderate or severe on the verbal categorical rating scale (VRS) and ≥4 on the numeric pain rating scale (NPRS)
* Surgical participants reporting pain at the surgical site that is moderate or severe on the VRS and ≥4 on the NPRS

Key Exclusion Criteria:

* Surgical participants:

  * History of previous surgery due to the same condition, except for procedures for which a previous surgery on the contra-lateral limb or organ is allowed
  * History of a prior surgical procedure in the same region of the body that resulted in any perioperative complications or that, in the opinion of the investigator or medical monitor, would preclude participation in the study
* History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Anaheim Clinical Trials, Anaheim, California
  - Trovare Clinical Research | Bakersfield, CA, Bakersfield, California
  - Mart Medical Research Group LLC, Miami, Florida
  - Mart Medical Research Group LLC, South Miami, Florida
  - Atlanta Center for Medical Research | Atlanta, GA, Atlanta, Georgia
  - Cypress Surgery Center, Wichita, Kansas
  - OrthoNebraska Hospital, Omaha, Nebraska
  - Center for Orthopaedic Reconstruction and Excellence, Jenks, Oklahoma
  - HD Research LLC | First Surgical Hospital, Bellaire, Texas
  - HD Research LLC | Legent Orthopedic Hospital, Carrollton, Texas
  - Renovatio Clinical, Houston, Texas
  - Futuro Clinical Trials, McAllen, Texas
  - South Texas Spine & Surgical Hospital, San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] McCoun J, Winkle P, Solanki D, Urban J, Bertoch T, Oswald J, Swisher MW, Taber LA, Healey T, Jazic I, Correll DJ, Negulescu PA, Bozic C, Weiner SG; VX-548-107 Study Team. Suzetrigine, a Non-Opioid NaV1.8 Inhibitor With Broad Applicability for Moderate-to-Severe Acute Pain: A Phase 3 Single-Arm Study for Surgical or Non-Surgical Acute Pain. J Pain Res. 2025 Mar 25;18:1569-1576. doi: 10.2147/JPR.S509144. eCollection 2025. PMID 40165940

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suzetrigine (SUZ)
Started | 258
Safety Set | 256 (Safety Set included all participants who received at least 1 dose of the study drug.)
Completed | 240
Not Completed | 18
Not completed — Withdrawal of consent (not due to AE) | 3
Not completed — Lost to Follow-up | 13
Not completed — Enrolled but not dosed | 2

BASELINE CHARACTERISTICS:
Population: Baseline data was analyzed based on the Full Analysis Set (FAS), defined as all participants who received at least 1 dose of study drug.
Groups:
- Suzetrigine (SUZ): Participants received SUZ 100 mg as first dose, followed by SUZ 50 mg q12h for 14 days or until pain resolves, whichever occurs first.
Arm/Group | Suzetrigine (SUZ)
Number analyzed (Participants) | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 108
  Not Hispanic or Latino | 148
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 214
  Black or African American | 34
  Asian | 3
  American Indian or Alaska Native | 3
  Native Hawaiian or other Pacific Islander | 1
  Multiracial | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Day 30
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Suzetrigine (SUZ)
Number analyzed (Participants) | 256
Participants
  Participants with TEAEs | 94
  Participants with SAEs | 2

2. Secondary Outcome: Percentage of Participants Reporting Good, Very Good, or Excellent on a Patient Global Assessment (PGA) Scale
Description: The PGA is a single-item assessment of patient perceptions of the method of pain control with the study drug and is evaluated on a 5-point Likert scale as: (poor, fair, good, very good or excellent). Percentage of participants who reported good, very good or excellent on the PGA scale was reported.
Time Frame: Day 14 or at Pain Resolution, whichever occurs first
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Suzetrigine (SUZ)
Number analyzed (Participants) | 256
percentage of participants | 83.2

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 30
Description: Safety Set included all participants who received at least 1 dose of study drug.
Arm/Group | Suzetrigine (SUZ)
All-Cause Mortality (participants affected / at risk) | 0/256
Serious Adverse Events (participants affected / at risk) | 2/256
Other Adverse Events (participants affected / at risk) | 18/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suzetrigine (SUZ) (N=256)
Cellulitis (Infections and infestations) | 1
Suicidal ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Suzetrigine (SUZ) (N=256)
Headache (Nervous system disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT05661734/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT05661734/SAP_001.pdf